CLINICAL TRIAL: NCT01283321
Title: RiaSTAP vs. Conventional Transfusion for Patients Undergoing Valve Replacement Surgery: RiaCT
Brief Title: RiaSTAP vs. Conventional Transfusion in Patients Having Heart Valve Surgery
Acronym: RiaCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding to complete total projected enrollment
Sponsor: Emory University (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Gautam Sreeram, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00036062; RiaCT 2010 (Other: Other)
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-05

CONDITIONS: Heart Valve Disease; Coronary Artery Disease
Keywords: Hemostasis; Cardiopulmonary bypass (heart-lung machine); Fibrinogen; platelet
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease | interventions — Fibrinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: RiaSTAP (Experimental): Human fibrinogen concentrate
  Interventions: Drug: Human fibrinogen concentrate
- Group B: apheresis platelets (Active Comparator): single apheresis unit
  Interventions: Other: apheresis platelets

INTERVENTIONS:
Drug: Human fibrinogen concentrate — 4 g IV once, within 30 minutes of ACT < 155 seconds, post CPB, with evidence of significant microvascular bleeding
  Other Names: RiaSTAP
  Arms: Group A: RiaSTAP
Other: apheresis platelets — A single apheresis platelet unit will be administered as an initial therapy within 30 minutes of ACT <155 seconds post CPB with evidence of significant microvascular bleeding.
  Arms: Group B: apheresis platelets

SUMMARY:
Heart surgery involving valve replacement often involves the use of the heart-lung machine for over 90 minutes, and bleeding tendency is frequently seen. Conventionally, platelet transfusion has been the primary therapy to treat bleeding after this type of procedure. More recently, perioperative supplementation of purified fibrinogen (RiaSTAP, CSL Behring) was shown to reduce bleeding and blood product use (plasma or platelets) after heart surgery. The objective of this trial is to demonstrate the clinical equivalency and economic utility of using fibrinogen concentrate, RiaSTAP for the mitigation of post-operative bleeding in patients in lieu of platelet transfusion.

Purified fibrinogen concentrate has been approved by FDA, and it has been used for the treatment of acute bleeding episodes in patients with low fibrinogen due to hereditary causes (e.g., afibrinogenemia). Compared to the transfusion of platelets which may be associated with volume overload, bacterial/viral infection, immunological effects and excess blood clotting, purified fibrinogen has several advantages. First, it contains no liquid plasma allowing for low volume infusion. Several viral inactivation/reduction steps are used to prepare the fibrinogen concentrate, increasing its viral safety. No antibodies or white blood cells are contained in the fibrinogen concentrate; therefore transfusion reactions are rare. Although platelet transfusion is widely used after heart surgery, there has been no randomized study to endorse this practice. In this study, patients undergoing heart valve replacement will be randomized to receive either platelet (1 unit) transfusion or fibrinogen concentrate (4g) after heparin anticoagulation is reversed. Subjects will be treated only if there is evidence of significant microvascular bleeding. Fifteen minutes after the initial treatment, subjects will be reevaluated for bleeding. If bleeding continues, subjects will be treated with blood transfusion per institutional standard of care.

The primary endpoints for this study are the hemostatic condition of the surgical field and 24-hour total of blood product transfusion.

DETAILED DESCRIPTION:
Platelet and plasma transfusion remain in the mainstay hemostatic therapy for perioperative bleeding. Several studies indicate that acquired fibrinogen deficiency can be the primary cause of bleeding after cardiac surgery. The aim of the study is to compare hematologica and transfusion profiles between the first-line fibrinogen replacement and platelet transfusion in post-cardiac surgical bleeding. In this prospective randomized, open-lable study, 20 adult patients undergoing valve replacement or repair, and fulfilling preset visual bleeding scale (0=excellent hemostasis; 1=oozing; 2=moderate bleeding; 3=severe bleeding from multiple bleeding sites) are randomized to 4 g of fibrinogen or 1 unit of apheresis platelet transfusion. After the initial randomized intervention, additional transfusions are given in the presence of bleeding (>200 ml/hour) according to the institutional practie as follows; 1 apheresis platelet unit if platelet count is less than 100 x 10^9 /L, 2 units of plasma if international normalized ratio is >1.6, or 10 units of cryoprecipitate if fibrinogen level is <200 mg/dL. Primary endpoints include hemostatic condition in the surgical field and 24-hour hemostatic product usage. Hematologica data, clinical outcome, and safety date are collected up to the 28th day postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age >17 and < 86 years
* Patients undergoing planned cardiopulmonary bypass (CPB) for:

  1. combined coronary artery bypass grafting and valve replacement/repair surgery
  2. single valve replacement surgery
  3. mitral valve repair surgery

  3. or double valve surgery (aortic and mitral)
* Presence of clinically relevant microvascular bleeding after protamine administration (hemostasis assessment score of 2-3)
* Patients should fulfill the following parameters prior to the study intervention:

  * Body temperature > 35.0°C
  * Blood pH > 7.2
  * Hb > 7.0 mg/dL
  * Activated clotting time (ACT) < 155 seconds
  * CPB time > 60 minutes

Exclusion Criteria:

* Replacement of aorta
* Planned valve replacement without median sternotomy
* Previous valve replacement surgery (previous coronary artery bypass graft (CABG) acceptable)
* History or suspicion of a congenital or acquired coagulation disorder such as hemophilia, von Willebrand disease, and liver disease
* Hemodialysis dependent renal failure
* Liver dysfunction (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) increased ≥ 2-fold above the upper limit of local laboratory normal ranges)
* Known allergy/anaphylaxis to fibrinogen concentrate or apheresis platelet units
* Clopidogrel administration within 5 days of surgery
* Coumadin (warfarin) administration within 5 days of surgery
* Participation in another clinical study in the 4 weeks preceding surgery
* Any indication that a potential subject did not comprehend the study restrictions, procedures, or consequences therein an informed consent cannot be convincingly given
* Life expectancy less than 48 hours

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Sreeram, MD, Principal Investigator — Emory University; Kenichi Tanaka, MD, MSc, Principal Investigator — University of Maryland
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tanaka KA, Egan K, Szlam F, Ogawa S, Roback JD, Sreeram G, Guyton RA, Chen EP. Transfusion and hematologic variables after fibrinogen or platelet transfusion in valve replacement surgery: preliminary data of purified lyophilized human fibrinogen concentrate versus conventional transfusion. Transfusion. 2014 Jan;54(1):109-18. doi: 10.1111/trf.12248. Epub 2013 May 30. PMID 23718572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started in February 2011 and the study was completed in May 2012. Subjects were recruited from Emory University. Fifty-one patients were approached after initial screening for eligibility, and 26 patients were consented.
Pre-assignment Details: Two subjects were excluded due to a change in surgical plans. Two subjects had low bleeding scores and were excluded.One subject had screening labs that were out of range for the study. One subject was treated using Dabigatran treatment. Total of six subjects that were excluded prior to randomization.
Period: Overall Study
Arm/Group | Group A: RiaSTAP | Group B: Apheresis Platelets
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 20 subjects were randomized after the screening visit/labs
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: RiaSTAP | Group B: Apheresis Platelets | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (5.3) | 66.1 (8.9) | 68.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Scores
Description: Bleeding scores are scored on a four-point scale. A visual assessment of surgical field was performed by the senior surgical staff as follows: 0 = excellent hemostasis (dry field), 1 = mild bleeding (oozing), 2 = moderate bleeding (controllable with applied pressure), and 3 = severe bleeding (multiple diffuse bleeding sites). If the visual bleeding scale was 2 to 3, the subjects were randomly assigned to a study intervention using a closed envelope method.
Time Frame: intra-operatively and up to 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: RiaSTAP | Group B: Apheresis Platelets
Number analyzed (Participants) | 10 | 10
units on a scale
  Intraoperative | 2.0 (0.0) | 2.1 (0.3)
  Postoperative | 1.0 (0.7) | 1.7 (0.8)

2. Secondary Outcome: Number of Participants in Whom Transfusion of Platelet Concentrate is Required During or After Surgery.
Time Frame: Operative period up to 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: RiaSTAP | Group B: Apheresis Platelets
Number analyzed (Participants) | 10 | 10
Participants | 4 | 10

3. Secondary Outcome: Volume (mL) of Fresh-frozen Plasma (FFP) Transfused-during Surgery and up to 24 Hours After Surgery
Time Frame: Operative period up to 60 minutes and up to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Group A: RiaSTAP | Group B: Apheresis Platelets
Number analyzed (Participants) | 10 | 10
ml | 0 [0 to 1300] | 650 [0 to 1300]

4. Secondary Outcome: Volume (mL) of Platelets Transfused- During Surgery and up to 24 Hours After Surgery
Time Frame: Operative period up to 60 minutes and up to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Group A: RiaSTAP | Group B: Apheresis Platelets
Number analyzed (Participants) | 10 | 10
ml | 0 [0 to 750] | 500 [250 to 1000]

5. Secondary Outcome: Median Blood Loss (mL) at 12 Hours After Surgery
Time Frame: From end of surgery to 12 hours after surgery
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Group A: RiaSTAP | Group B: Apheresis Platelets
Number analyzed (Participants) | 10 | 10
ml | 925 [500 to 1693] | 1315 [653 to 2965]

ADVERSE EVENTS:
Time Frame: Reported adverse events (AEs) include events starting during the surgery (intraoperative) and on and before 30 days after surgery (post-operative).
Arm/Group | Group A: RiaSTAP | Group B: Apheresis Platelets
Serious Adverse Events (participants affected / at risk) | 1/10 | 6/10
Other Adverse Events (participants affected / at risk) | 3/10 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: RiaSTAP (N=10) | Group B: Apheresis Platelets (N=10)
Atrial Fibrillation (Cardiac disorders) | 0 | 2
Excessive mediastinal bleeding (Injury, poisoning and procedural complications) | 1 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: RiaSTAP (N=10) | Group B: Apheresis Platelets (N=10)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 5

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No